CLINICAL TRIAL: NCT02871024
Title: Efficacy of Polymyxin B Hemoperfusion on Severe Sepsis Secondary to Pneumonia or Urinary Tract Infection: A Single-arm Clinical Trial
Brief Title: Efficacy of Polymyxin B Hemoperfusion on Severe Sepsis Secondary to Pneumonia or Urinary Tract Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Ms. Ying Ting Chao, Sheng-Yuan Ruan MD, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201411023RIPB
Record Dates: First submitted 2016-08-04; First posted 2016-08-18 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Sepsis
Keywords: Polymyxin B; Pneumonia; Sepsis; Urinary tract infection
MeSH Terms: conditions — Sepsis; Pneumonia; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): Usual care with two sessions of 2-hour hemoperfusion with Toraymyxin in 24 hours apart
  Interventions: Device: Toraymyxin

INTERVENTIONS:
Device: Toraymyxin — Toraymyxin is an extracorporeal hemoperfusion device designed to reduce blood endotoxin levels in sepsis

SUMMARY:
Toraymyxin is an extracorporeal hemoperfusion cartridge containing Polymyxin B-immobilized fiber column designed to reduce blood endotoxin levels in sepsis. Meta-analysis of randomized trials showed that polymyxin B hemoperfusion significantly reduced the mortality of severe sepsis; however, the evidence was mainly contributed by the studies of abdominal sepsis. The data about using polymyxin B hemoperfusion to treat non-abdominal sepsis remain very limited. Investigators designed a clinical trial to evaluate the efficacy of polymyxin B hemoperfusion on treating non-abdominal severe sepsis. The study hypothesis is that removal of endotoxin by polymyxin B hemoperfusion in patients with pneumonia or urinary tract infection (UTI)-related severe sepsis will attenuate sepsis associated microcirculation failure and result in early reversal of shock and less extent of end-organ damage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with septic shock defined by the third international consensus definitions for sepsis and septic shock
2. Newly diagnosed pneumonia or urinary tract infection (UTI) defined as the following:

   2-1. Pneumonia is defined by a new infiltrate on chest radiograph and the presence of one or several of the following signs or symptoms: cough, sputum production, dyspnea, core body temperature ≥ 38.0°C, auscultatory findings of abnormal breath sounds and rales and leukocyte count > 10000 or < 4000/L.

   2-2. UTI is defined by at least one clinical symptom (core body temperature ≥38.0°C, urinary urgency, polyuria, dysuria, suprapubic pain, flank pain, costovertebral angle tenderness, nausea and vomiting) and one urinary criterion (pyuria >20 leukocytes/μL).
3. Hyperlactatemia (>2 mmol/L)
4. Endotoxin activity assay (EAA) ≥ 0.5 units.

Exclusion Criteria:

1. Shock persisted >12 hours before screening
2. Mechanical ventilation >21 days
3. Uncontrolled hemorrhage
4. Thrombocytopenia (platelet count < 30,000 cells/mm3)
5. Leukopenia (leukocyte count < 1500 cells/mm3)
6. Suspected allergy to polymyxin
7. Females with pregnancy
8. Terminal cancer or organ failure with life expectancy less than 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08; Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Reversal of sepsis-associated circulatory failure | Day 7
  Comparison of the proportion of subjects free from vasopressor on Day 7 between the intervention group and historical control group.

SECONDARY OUTCOMES:
Lactate clearance of survived subjects | Day 3
  Comparison of lactate clearance between the intervention group and historical control group. Lactate clearance = (initial lactate level - subsequent lactate level) / (initial lactate level)
Change of endotoxin levels (Endotoxin Activity Assay) | Day 3
  Change of endotoxin levels after the intervention
Change of Sequential Organ Failure Assessment (SOFA) score | Day 7
  Comparison of SOFA score between the intervention group and historical control group.
Vasopressor-free days | 7 days
  Comparison of vasopressor-free days in 7 days between the intervention group and historical control group.
28-day all-cause mortality | 28 days
  Comparison of 28-day all-cause mortality between the intervention group and historical control group.
Catheter-related complications | 3 days
  Comparison of the proportion of the cases with catheter-related complications between the intervention group and historical control group.
Thrombocytopenia (<25,000/μL) | 3 days
  Comparison of the proportion of the cases with thrombocytopenia (<25,000/μL) between the intervention group and historical control group.
Cases with major bleeding needed transfusion with packed red blood cells > 2 units/day | 3 days
  Comparison of the proportion of the cases with major bleeding between the intervention group and historical control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Yuan Ruan, MD, Principal Investigator — Natioanl Taiwan University Hospital, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided